CLINICAL TRIAL: NCT05482646
Title: Tai Chi Versus Conventional Exercise to Alleviate Depressive Symptoms in Older Insomniacs: A Three-arm Randomized Controlled Trial
Brief Title: Tai Chi Versus Conventional Exercise to Alleviate Depression in Insomniacs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Parco M. Siu, PhD, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TaiChiTrialHKU2020
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Depressive Symptoms; Chronic Insomnia
Keywords: Exercise; Tai Chi; Elderly; Depression; Insomnia
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders; Motor Activity | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi (Experimental): This group will perform 3 months of Tai Chi training
  Interventions: Behavioral: Tai Chi
- Conventional exercise (Active Comparator): This group will perform 3 months of conventional exercise training
  Interventions: Behavioral: Conventional exercise
- Health Education Control (Other): This group will participate in a 3-month health education program
  Interventions: Behavioral: Health Education Control

INTERVENTIONS:
Behavioral: Tai Chi — The Tai Chi intervention will be prescribed as a 3-month program with two 1.5-h sessions weekly instructed by qualified Tai Chi instructors.
  Arms: Tai Chi
Behavioral: Conventional exercise — The conventional exercise intervention will be prescribed as a 3-month program with two 1.5-h sessions of generic fitness training weekly instructed by qualified instructors.
  Arms: Conventional exercise
Behavioral: Health Education Control — Participants in the control group will participate in a health education program delivered by research personnel.
  Arms: Health Education Control

SUMMARY:
This study aims to examine the effectiveness of Tai Chi and conventional exercise in alleviating depressive symptoms in older insomniacs.

DETAILED DESCRIPTION:
Chinese community-dwelling older adults with mild-to-moderate depressive symptoms and chronic insomnia will be recruited.

Eligible participants will be randomized to health education control, Tai Chi or conventional exercise interventions on a 1:1:1 basis after baseline assessment.

All interventions will last for 3 months. Outcomes will be assessed at baseline, at 3 months and at 6 months after the completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* Can communicate using Cantonese or Mandarin
* with mild-to-moderate depressive symptoms (HADS-depression score ≥8/21 and PHQ- 9 score ≤14/27)
* Fulfil the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for chronic insomnia including difficulties in initiating or maintaining sleep, early morning awakening with complaint of significant distress or impairment of daytime functioning, sleep difficulty occurring at least three nights per week and present for at least 3 months.

Exclusion Criteria:

* Somatic condition that prevents participation in tai chi or exercise
* Regular moderate-to-vigorous intensity exercise or mind-body training such as tai chi, yoga, qigong or meditation in the past 3 months
* Any form (or combination) of exercises amounting to 180 minutes per week in the past 3 months
* Dementia
* Diagnosis with schizophrenia or other psychotic disorders, bipolar disorders or alcohol/substance use/abuse
* Current usage or planning to use potentially confounding treatments, including herbal supplementations (e.g., St. John's Wort), acupuncture treatment, cognitive behavioral therapy or other psychotherapy, mind-body intervention (e.g., mindfulness training and muscle relaxation training) or muscle relaxants such as carisoprodol, cyclobenzaprine, diazepam
* Current suicidal or self-injurious potential that requires immediate clinical follow-up.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale - Depression | 3 months (post-intervention)
  The depression score of the Hospital Anxiety and Depression Scale (HADS-D) will be used to evaluate the severity of depressive symptoms. This consists of a seven-item questionnaire with an overall score ranging from 0 to 21. Higher scores are indicative of more severe depressive symptoms.
Hospital Anxiety and Depression Scale - Depression | 9 months (6 months post-intervention follow-up)
  The depression score of the Hospital Anxiety and Depression Scale (HADS-D) will be used to evaluate the severity of depressive symptoms. This consists of a seven-item questionnaire with an overall score ranging from 0 to 21. Higher scores are indicative of more severe depressive symptoms.

SECONDARY OUTCOMES:
Insomnia severity index | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  The Insomnia Severity Index (ISI) will be used to assess perceived insomnia severity. It consists of a seven-item questionnaire with each item being rated from 0 to 4 on a Likert scale (total score range 0-28). Higher scores are representative of a more severe perception of insomnia.
Pittsburgh Sleep Quality Index | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess subjective sleep quality. It consists of a 19-item questionnaire designed to measure sleep quality and disturbance. The 19 items are grouped into 7 components, and each component yields a score ranging from 0 to 3, with 3 indicating the greatest sleep dysfunction. The total score of the PSQI ranges from 0 to 21, with higher scores indicating worse sleep quality.
Patient Health Questionnaire | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  The Patient Health Questionnaire (PHQ-9) will be used to assess the severity of depression. The questionnaire is composed of 9 items, with each item being rated from 0 to 3. The PHQ-9 has a total score ranging from 0 to 27, with higher scores suggesting higher depressive symptom severity.
General Anxiety Disorder Scale | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  The General Anxiety Disorder Scale (GAD-7) will be used to assess the severity of anxiety. The GAD-7 is composed of 7 items, each being rated from 0 to 3 and with a total score range of 0-21. Higher scores are representative of greater anxiety symptoms.
Hospital Anxiety and Depression Scale - Anxiety | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  The anxiety score of the Hospital Anxiety and Depression Scale (HADS-A) will be used to assess the severity of anxiety symptoms. The HADS-A consists of a seven-item questionnaire with an overall score ranging from 0 to 21. Higher scores are indicative of greater anxiety symptoms.
Medication usage | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  The use of medications will be recorded.
The 12-item Short Form Survey | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  The 12-item Short Form Survey (SF-12) will be used to measure health-related quality of life. It consists of 12 items that are aggregated to form 2 summary scores: mental component score (MCS) and physical component score (PCS). Both MCS and PCS have a scoring range of 0 to 100, with higher scores indicating better mental and physical functioning.
Short Physical Performance Battery | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  The Short Physical Performance Battery (SPPB) will be used to assess physical function and balancing performance. The SPPB involves repeated timed chair stands and a 4-meter walk to measure gait speed. Scores ranging from 1 to 4 are assigned based on test results, with higher scores indicating better physical function and balance.
Sleep efficiency through actigraph | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  Sleep efficiency will be objectively evaluated by means of an actigraph. Sleep efficiency is the ratio between the time spent asleep and the total time spent in bed (expressed as %). Higher rates are indicative of healthier sleep patterns.
Sleep efficiency through sleep diary | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  Sleep efficiency will be subjectively evaluated by means of a sleep diary. Sleep efficiency is the ratio between the time spent asleep and the total time spent in bed (expressed as %). Higher rates are indicative of healthier sleep patterns.
Wake time after sleep onset through actigraph | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  Wake time after sleep onset will be objectively measured by means of an actigraph. It represents the total number of minutes that a person is awake after having initially fallen asleep (expressed as minutes). Higher values are indicative of more severe sleep problems.
Wake time after sleep onset through sleep diary | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  Wake time after sleep onset will be subjectively measured by means of a sleep diary. It represents the total number of minutes that a person is awake after having initially fallen asleep (expressed as minutes). Higher values are indicative of more severe sleep problems.
Number of awakenings through actigraph | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  The number of awakenings will be objectively measured by means of an actigraph. It represents the total number of times that the participant woke up throughout the night (expressed as N). Higher values indicate worse sleep patterns.
Number of awakenings through sleep diary | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  The number of awakenings will be subjectively measured by means of a sleep diary. It represents the total number of times that the participant woke up throughout the night (expressed as N). Higher values indicate worse sleep patterns.
Sleep onset latency through actigraph | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  Sleep onset latency will be objectively measured by means of an actigraph. It represents the time that it takes for a participant to fall asleep and is expressed in minutes. Higher values are indicative of worse sleep patterns.
Sleep onset latency through sleep diary | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  Sleep onset latency will be subjectively measured by means of a sleep diary. It represents the time that it takes for a participant to fall asleep and is expressed in minutes. Higher values are indicative of worse sleep patterns.
Average awake time through actigraph | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  Average awake time will be objectively measured by means of an actigraph. It is expressed as wake time after sleep onset divided by the number of awakenings, and is expressed in minutes. Higher values represent worse sleep patterns.
Average awake time through sleep diary | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  Average awake time will be subjectively measured by means of a sleep diary. It is expressed as wake time after sleep onset divided by the number of awakenings, and is expressed in minutes. Higher values represent worse sleep patterns.
Total sleep time through actigraph | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  Total sleep time will be objectively measured by means of an actigraph. It represents the total number of minutes spent asleep during the sleep period (expressed as minutes). Higher values are indicative of healthier sleep patterns.
Total sleep time through sleep diary | 3 months (post-intervention) and 9 months (6 months post-intervention follow-up)
  Total sleep time will be subjectively measured by means of a sleep diary. It represents the total number of minutes spent asleep during the sleep period (expressed as minutes). Higher values are indicative of healthier sleep patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Parco M Siu, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- LKS Faculty of Medicine, HKU, Hong Kong, Hong Kong